CLINICAL TRIAL: NCT06170775
Title: Sodiumhexametaphosphate Versus MTA as Pulp Capping Material for Primary Teeth ( Randomized Clinical Trial)
Brief Title: Sodiumhexametaphosphate as Pulp Capping Material for Primary Teeth
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Minia University (Other)
Responsible Party: Principal Investigator, Mahmoud Ahmed Mahmoud, Lecturer, Minia University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1290
Record Dates: First submitted 2023-12-06; First posted 2023-12-14 (Actual); Last update posted 2023-12-14 (Actual); Status verified 2023-12

CONDITIONS: Pulp Disease, Dental
MeSH Terms: conditions — Dental Pulp Diseases | interventions — Pemetrexed

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sodiumhexametaphosphate (Experimental)
  Interventions: Other: Pulp therapy; Drug: Sodiumhexametaphosphate
- MTA (Active Comparator)
  Interventions: Other: Pulp therapy; Other: MTA

INTERVENTIONS:
Other: Pulp therapy — Pulp capping material
Drug: Sodiumhexametaphosphate — Sodiumhexametaphosphate
  Arms: Sodiumhexametaphosphate
Other: MTA — MTA
  Arms: MTA

SUMMARY:
Sodiumhexametaphosphate will be tested as pulp capping material in comparison to MTA for primary teeth pulp therapy

ELIGIBILITY:
Inclusion Criteria:

* physical healthy children
* cooperative children
* primary molar with deep carious lesion
* absence of pain or transient momentary pain

Exclusion Criteria:

* Uncooperative children
* children with systemic disorders
* periapical lesions
* sever pain

Ages: 4 Years to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 100 (Estimated)
Dates: Start 2023-12-20 (Estimated); Primary Completion 2024-12-20 (Estimated); Study Completion 2025-01-20 (Estimated)

PRIMARY OUTCOMES:
Clinical success | One year
  Absence of pain, swelling and sinus tract
Radiographic success | One year
  Absence of periapical lesions, internal or external root resorption